CLINICAL TRIAL: NCT06036966
Title: The Efficacy and Safety of Hetrombopag in Primary Prevention of Thrombocytopenia Induced by the Niraparib Maintenance in Advanced Ovarian Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-764-02
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Thrombocytopenia
Keywords: Niraparib; Hetrombopag; Primary prevention
MeSH Terms: conditions — Thrombocytopenia | interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag (Experimental): single-arm
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — All the enrolled 34 patients will be given hetrombopag 5mg per day for 8 weeks when they start to take Niraparib as maintenance therapy

SUMMARY:
Niraparib brings a better prognosis to those with advanced ovarian cancer and has been approved by the Food and Drug Administration（FDA ）and National Medical Products Administration（NMPA）as one of the maintenance therapies for the advanced ovarian cancer patients. Thrombocytopenia is one of the adverse effects of Niraparib, with a 61% overall incidence and 34% of the grade 3~4 incidence. Thrombocytopenia may cause suspension or dose reduction of Niraparib which will affect the therapeutic effect of the drug.

At present, the drugs recommended by the guidelines for the treatment of thrombocytopenia are recombinant thrombopoietin (rhTPO), recombinant interleukin 11 (rhIL-11), TPO receptor agonist (TPO-RA). Hetrombopag is one of the TPO-RA, which is recommended by the Chinese expert consensus to cure the thrombocytopenia caused by poly adenosinediphosphate ribose polymerase（PARP） inhibitors, including Niraparib. However, is it effective when it is used as the primary prevention during the maintenance therapy of Niraparib? This single-arm study aims to explore the efficacy and safety of hetrombopag for the prevention of thrombocytopenia caused by Niraparib maintenance therapy in advanced ovarian cancer patients. 34 patients will be recruited and they will take hetrombopag 5mg per day for 8 weeks when they initiate the maintenance therapy with Niraparib. The primary endpoint of this study is the rate of thrombocytopenia according to Common Terminology Criteria for Adverse Events 5.0（CTCAE5.0）.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Ovarian cancer patients using niraparib as maintenance therapy;
3. Estimated survival≥ 12 weeks;
4. Eastern Cooperative Oncology Group Physical Score(ECOG PS) : 0-2;
5. Adequate function of organs:

(1) Platelet count 100-300*109/L, neutrophil count≥2.0*109/L, hemoglobin 100-150g/L; (2) Renal function: Cr≤1.5 upper limit of normal（ULN）; (3) Endogenous creatinine clearance (Ccr) ≥ 55 ml/min; (4) Liver function: total bilirubin ≤1.5 upper limit of normal（ULN）; (5) Alanine aminotransferase（ALT）and aspartate aminotransferase（AST）≤3 upper limit of normal（ULN）; (6) Coagulation function: PT≤1.5 upper limit of normal（ULN）; 6. No serious complications (including active gastrointestinal bleeding, perforation, jaundice, gastrointestinal obstruction, non-cancerous fever> 38℃)

Exclusion Criteria:

1. Patients with the following hematopoietic system diseases: leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma and myelodysplastic syndrome, etc;
2. Thrombocytopenia caused by non-anti-tumor therapy within 6 months before screening, including chronic liver disease, hypersplenism, infection and bleeding, etc;
3. Imaging examination shows bone marrow invasion or bone marrow metastasis, such as Positron Emission Computed Tomography（PET-CT）, Magnetic Resonance Imaging（MRI）or nuclear scan;
4. Patients with antiphospholipid syndrome;
5. Platelet transfusion or used TPO-RA, rhTPO and other platelet-raising drugs within 3 days before screening;
6. Patients with known or expected hypersensitivity or intolerance to the active ingredient or excipients of Hetrombopag

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-09-16 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
efficacy of hetrombopag | from the date of recruitment to the time of 12 weeks
  incidence of thrombocytopenia according to Common Terminology Criteria for Adverse Events 5.0(CTCAE5.0)

SECONDARY OUTCOMES:
incidence of Niraparib suspension | from the date of recruitment to the time of 12 weeks
  incidence of Niraparib suspension due to thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No